CLINICAL TRIAL: NCT06379516
Title: Comprehensive Process Validation of Dermatological Wound Creation Techniques: A Study Evaluating Methodology Standardization for Assessment of Treatment Efficacy in Controlled Skin Damage
Brief Title: Process Validation in Dermatology: Assessing Wound Creation Methods and Treatment Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Principal Investigator, Maheshvari Patel, Principal Investigator - Director (Operations), NovoBliss Research Pvt Ltd
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NB240004-NB-V
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Validation of the Process of Wound Creation and Evaluation
MeSH Terms: interventions — Coconut Oil

STUDY DESIGN:
Intervention Model Description: Proof of science/concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moisturising Cream A (Active Comparator)
  Interventions: Other: Moisturising Cream (5%)
- Moisturising Cream B (Active Comparator)
  Interventions: Other: Moisturising Cream (10%)
- Test Oil (Placebo Comparator)
  Interventions: Other: Coconut Oil
- Untreated (No Intervention)

INTERVENTIONS:
Other: Moisturising Cream (5%) — This intervention is a moisturiging cream of concentration 5% for topical application to the respective test sites.
  Arms: Moisturising Cream A
Other: Moisturising Cream (10%) — This intervention is a moisturiging cream of concentration 10% for topical application to the respective test sites.
  Arms: Moisturising Cream B
Other: Coconut Oil — This intervention is a 100% pure coconut oil product (Parachute Pure Coconut Oil) for topical application to the respective test sites.
  Arms: Test Oil

SUMMARY:
The primary objective of this study is to validate controlled methods of wound, including 1%w/v SLS, 3%w/v SLS, and 24-24 times tape stripping, on the forearms of subjects.

The study aims to standardize the procedures for creating wounds and systematically evaluate the effects of these methods on various skin parameters.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is aged between 18 and 55 years (both inclusive) at the time of informed consent.
2. The subject is a healthy adult male, or a non-pregnant, non-lactating, healthy adult female.
3. No previous history of adverse skin conditions, and not under any medication likely to interfere with the results.
4. The subject, if female, has a self-reported negative urine pregnancy test.
5. The subject is in a good general health as determined from recent medical history.
6. The subject has willingness and ability to adhere to study directions, and agrees not to use any other skin creams, lotions, serums, etc. at the application sites, except for the specified test products, and return for all specified visits.
7. The subject possesses the ability to comprehend and provide written informed consent for participation in the study.

Exclusion Criteria:

1. The subject is currently pregnant/lactating or is planning to become pregnant during the study period.
2. The subject has a history of allergies or specific allergic reactions upon using dermatological/cosmetic products.
3. The subject is currently enrolled in an active investigational study or has participated in an investigational study within 30 days prior to enrolment.
4. The subject suffers from any active clinically significant disease or any condition that according to the investigator's discretion warrants exclusion from the study.
5. The subject is taking or has taken a medication which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Trans Epidermal Water Loss (TEWL) | Days -02, -01, 01, 02, 05, 08, 28
  Using the Tewameter® TM Hex
Skin hydration | Days -02, -01, 01, 02, 05, 08, 28
  Using the Corneometer® CM 825
Skin surface topography | Days -02, -01, 01, 02, 05, 08, 28
  Assessment of skin smoothness, scaliness, roughness, wrinkles using the Visioscan® VC 20plus.

SECONDARY OUTCOMES:
Dermatological Assessment | Days -02, -01, 01, 02, 05, 08, 28
  Visual dermatological evaluation of the skin using the Draize scale where 0 indicates no reactions and 4 indicates severe reactions

CONTACTS AND LOCATIONS:
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No